CLINICAL TRIAL: NCT01745536
Title: "Impact of a Closed System in Donor Oocyte Vitrification"
Brief Title: Closed Vitrification of Oocytes
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: NO RECRUITMENT
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Responsible Party: Principal Investigator, Ana Cobo, Cryo-biology Unit director at IVI Valencia, Spain, Instituto Valenciano de Infertilidad, IVI VALENCIA
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 1206-C-104-AC; Clinical Trials.gov (Registry Identifier: Clinical Trials.gov)
Record Dates: First submitted 2012-11-29; First posted 2012-12-10 (Estimated); Last update posted 2016-03-08 (Estimated); Status verified 2016-03

CONDITIONS: Infertility
Keywords: Oocyte vitrification; survival rate; egg banking; ovum donation
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitrified oocytes using closed Cryotop® (Experimental): Oocytes are vitrified/stored using a closed device
  Interventions: Procedure: Oocytes are vitrified/stored using a closed device
- Vitrified oocytes using open Cryotop® (Active Comparator): Oocytes are vitrified/stored using an open device
  Interventions: Procedure: Oocytes are vitrified/stored using an open device

INTERVENTIONS:
Procedure: Oocytes are vitrified/stored using a closed device — Vitrification will be carried out using a modification of the current device (Cryotop®), thus providing air tight sealing. Closed systems are devices that are hermetically sealed before vitrification and remain sealed during storage.
  Arms: Vitrified oocytes using closed Cryotop®
Procedure: Oocytes are vitrified/stored using an open device — The vitrification process takes place through direct contact with liquid nitrogen. The system has an external straw to protect the samples during storage, but the device is not hermetically sealed.
  Arms: Vitrified oocytes using open Cryotop®

SUMMARY:
This study is aimed to evaluate the use of a closed device for storage of vitrified oocytes.

DETAILED DESCRIPTION:
The Cryotop method for oocyte vitrification is classified as "open system", which means that it requires direct contact with liquid nitrogen during the vitrification process. The system has an external straw to protect the samples during storage, but the device is not hermetically sealed. Instead closed systems are devices that are hermetically sealed before vitrification and remain sealed during storage. Open systems have proven highly effective in achieving similar outcomes with vitrified oocytes compared to those achieved with fresh ones. On the contrary, closed systems have failed to be as effective as open ones when used for oocyte vitrification. Although open systems have proven to be highly efficient, where many other methods have failed, they have been related to a theoretical risk of contamination due to direct contact with liquid nitrogen. Though to date there have been no reported cases of transmission of disease after cryo-transfers either for slow freezing or vitrification, some European countries prohibit the use of open systems for vitrification. In this study, we will evaluate the results after the donor oocyte vitrification, using a modification of a current device (Cryotop®), which makes it capable of being hermetically sealed. The current study is a prospective randomized trial aimed to assess the outcome of ovum donation cycles conducted with vitrified oocytes using the closed device versus oocytes vitrified using the traditional open device.

ELIGIBILITY:
Inclusion Criteria:

Donors:

* < 35 years old
* Normal physical and gynecological examinations
* No family history of hereditary or chromosomal diseases.
* Normal karyotype
* Negative screening for sexually transmitted diseases.

Oocyte recipients:

* Oocyte recipients < 50 years old
* Body mass index < 30
* < 2 previous IVF failures
* No severe male factor
* No recurrent miscarriage
* No hidrosalpinx
* No myoma
* No adenomyosis
* No AMH alterations

Exclusion Criteria:

Donors and recipients not meeting inclusion criteria

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2012-11; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Survival after oocyte vitrification using the closed device Cryotop® | >2 hours
  Survival will be evaluated morphologically two hours after warming.

SECONDARY OUTCOMES:
Embryo development | From thawing and until pregnancy outcome (0-9 months)

CONTACTS AND LOCATIONS:
Overall Officials: Ana Cobo, PhD, Principal Investigator — IVI Valencia
Locations (2):
- Spain (2):
  - Ivi Valencia, Valencia, Valencia
  - IVI Valencia, Valencia